CLINICAL TRIAL: NCT07340086
Title: Assessment of Emotional and Empathic Involvement During Simulation-Based Communication Training in Nursing Students
Brief Title: Mobilization of Emotions and Empathy During Communication Training in Nursing Students
Acronym: AEI-Sim
Status: Active, not recruiting | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: Pontifical Catholic University of Argentina (Other)
Responsible Party: Sponsor
Other Study IDs: AEI-Sim-2025-01
Record Dates: First submitted 2025-12-16; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Education Nursing; Communication Skills; Ethics Education; Empathy; Simulation Based Learning
Keywords: Nursing; Education; Communication skills; Simulation; Ethics; Empathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Effective communication in healthcare is vital for patient satisfaction, safety, outcomes, and ethical practice, supporting shared decision-making and informed consent. Simulation-based training is widely used to strengthen communication skills and foster empathy through emotionally engaging experiences.

This is a pilot study aimed (1) to assess changes in emotional state and empathy in nursing students after a simulation-based workshop (SBW) on delivering bad news, and (2) to evaluate the sensitivity of standardized scales in detecting these changes.

DETAILED DESCRIPTION:
In this observational, longitudinal study, fourth-year nursing students (Pontifical Catholic University of Argentina - Pontificia Universidad Católica Argentina, Buenos Aires) attended a curricular six-hour SBW divided into three sessions. In Session 1, students discussed the SPIKE protocol for communication of bad news, and a clinical case, completing a baseline Positive and Negative Affect Schedule (PANAS). In Session 2, students performed role-plays with simulated patients (SPs), immediately after which the students registered their emotional reflections (ER), completing the Jefferson Scale of Empathy for Health Professionals (JSE-HP), the Jefferson Scale of Patient Perceptions of Physician Empathy (JSPPPE) adapted for nursing communication and repeated PANAS; instructors and SPs also completed JSPPPE. In Session 3, students participated in debriefing and repeated ER, JSE-HP and JSPPPE.

PANAS is a mood scale with 20 items, 10 positive (PA) and 10 negative (NA). High PA means "enthusiastic and motivated"; low PA means "lethargic and sad." High NA means "angry and disgusted"; low NA means "calm and serene." JSE-HP is a 20-item empathy scale for healthcare settings. It measures how well a healthcare professional understands and communicates a patient's perspective. The 7-point Likert scale ranges from 20 to 140.

JSPPE is a 5-item patient-completed empathy scale for healthcare professionals. It uses a 1-to-7 Likert scale to assess understanding, concern, and perspective-taking. Max score: 35 points.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students of the 4th year

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fourth-year nursing students who conducted a simulation-based workshop as part of their communication training curriculum.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes of emotions after the simulation-based workshop on communication of bad news | The PANAS score was completed after sessions 1 (baseline, day 0), 2 (simulation, 1 week after day 0), and 3 (debriefing, 2 weeks after day 0). Baseline day: August 1, 2025. Session 2: August 8, 2025. Session 3: August 15, 2025.
  Questionnaires from the PANAS were completed by the participants.

SECONDARY OUTCOMES:
Changes of empathy during a simulation-based workshop on communication of bad news measured by Jefferson Scale of Empathy. | Students completed the JSE questionnaire after sessions two and three of the three-stage, simulation-based workshop on communicating bad news. Session two took place on August 8, 2025, and session three took place on August 15, 2025.
  Participants recorded their changes by filling out the Health Professions Version of the Jefferson Scale of Empathy (JSE), which was adapted for nursing communication.
Changes of perceived empathy after participating in a simulation-based workshop on communication of bad news measured by Jefferson Scale of Patient Perceptions of Physician Empathy | Complete the JSPPPE after sessions two and three, or the simulation and debriefing days (August 8 and 15, 2025), of the three-stage, simulation-based workshop on communicating bad news.
  Self-perceived empathy was scored during the communication of bad news using the Jefferson Scale of Patient Perceptions of Physician Empathy (JSPPPE).

OTHER OUTCOMES:
Changes in self-perceived emotions while executing the simulation-based workshop on communication of bad news | Records were taken after Session 2 (Simulation Day, August 8, 2025) and Session 3 (Debriefing Day, August 15, 2025).
  Participants recorded their self-perceived emotions (emotional reflections) by writing about their feelings, emotions, and sensations in a logbook.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Martinato, PhD, Study Director — University of Padova
Locations (1):
- Pontifical Catholic University of Argentina, Buenos Aires, Argentina